CLINICAL TRIAL: NCT03232593
Title: Post-Marketing Surveillance of Tecentriq in MFDS-Approved Indication(s)
Brief Title: A Study of Atezolizumab (Tecentriq®) in Ministry of Food and Drug Safety (MFDS)-Approved Indication(s)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML39313
Record Dates: First submitted 2017-07-26; First posted 2017-07-28 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Urothelial Carcinoma; Carcinoma, Non-Small Cell Lung; Small Cell Lung Carcinoma; Triple Negative Breast Carcinoma; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Triple Negative Breast Neoplasms; Carcinoma, Hepatocellular | interventions — atezolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Participants who Receive Atezolizumab: Participants who are administered with atezolizumab as per the local label and standard of care at physician's discretion will be observed for approximately 6 years.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Participants will receive atezolizumab as per the local label and standard of care at physician's discretion.
  Other Names: Tecentriq

SUMMARY:
This Phase 4, prospective, multicenter, non-interventional, regulatory post-marketing surveillance study will collect information on the the safety and effectiveness of atezolizumab under the clinical practice, and update the drug label approved by the MFDS in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are administered with atezolizumab for the locally approved indications

Exclusion Criteria:

* Participants with a known hypersensitivity to atezolizumab or to any of the excipients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who are administered with atezolizumab at physician's discretion will be enrolled for the study.
Sampling Method: Non-Probability Sample
Enrollment: 1758 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) and Serious AEs (SAEs) | Approximately 6 years

SECONDARY OUTCOMES:
Percentage of Participants With Complete Response (CR) Assessed per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Approximately 6 years
Percentage of Participants With Partial Response (PR) Assessed per RECIST 1.1 | Approximately 6 years
Percentage of Participants With Stable Disease (SD) Assessed per RECIST 1.1 | Approximately 6 years
Percentage of Participants With Progressive Disease (PD) Assessed per RECIST 1.1 | Approximately 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (56):
- South Korea (56):
  - Dongnam Inst.of Radiological & Medical Sciences, Busan
  - Inje University Busan Paik Hospital, Busan
  - Inje university Haeundae Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Donga Uni Medical Center; Pulmonary, Busan
  - Pusan University Hospital, Busan
  - Pusan University Hospital; Hemato-oncology, Busan
  - Kyungpook National University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Hospital; Pulmonology, Daegu
  - Konyang University Hospital, Daejeon
  - Hallym University Medical Center Chuncheon Sacred Heart Hospital, Gangwon-do
  - Yonsei University Wonju Severance Christian Hospital, Gangwon-do
  - Gangneung Asan Hospital, Gangwon-do
  - Uijeongbu St. Mary's Hospital, Gyeonggi-do
  - CHA Bundang Medical Center, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Gyeonggi-do
  - Soonchunhyang University Bucheon Hospital, Gyeonggi-do
  - Bucheon St Mary's hospital, Gyeonggi-do
  - Korea University Ansan Hospital, Gyeonggi-do
  - St. Vincent's Hospital, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Gyeongsangnam-do
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si
  - Chonbuk National University Hospital, Jeollabuk-do
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Wonkwang University School of Medicine & Hospital, Jeonlabuk-do
  - Korea Cancer Center Hospital of Korea Institute of Radiological and Medical Sciences, Seoul
  - Korea University Anam Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Eunpyeong St. Mary's Hoapital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Soonchunhyang University Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Gangdong Kyung Hee University Hospital, Seoul
  - VHS Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
  - ChungAng University Hospital, Seoul
  - Borame Medical Center, Seoul
  - Yeouido St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Severance Hospital, Yonsei University Health System; Oncology, Seoul
  - Samsung Medical Centre; Division of Hematology/Oncology, Seoul
  - Ewha Womans University Mokdong Hospital; Urology, Seoul
  - Korea Uni Anam Hospital; Internal Medicine, Seoul
  - SoonChunHyang University Hospital Seoul, Seoul
  - Ulsan University Hosiptal, Ulsan
  - Ulsan University Hospital, Ulsan
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
  - Pusan National University Yangsan Hospital; hemato-oncology, Yangsan